CLINICAL TRIAL: NCT05792371
Title: The Role of Endothelial Cell-mediated Type H Vessel Formation in Induced Membrane-enhanced Bone Union of Patients With Critical Size Bone Defect
Brief Title: The Role of Type H Vessel Formation in Induced Membrane of Patients With Critical Size Bone Defect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 202201532B0A3
Record Dates: First submitted 2023-02-15; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-01

CONDITIONS: Bone Injury
Keywords: Induced membrane; Bone healing; Type H vessel
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with induced membrane (Experimental): operation of stage I and II
  Interventions: Procedure: induced membrane technique
- without induced membrane (Experimental): only stage II
  Interventions: Procedure: Bone graft (Stage II of IMT)

INTERVENTIONS:
Procedure: induced membrane technique — Masquelet technique, also called an induced membrane technique (IMT), was first introduced to treat critical size bone defect up to 25 cm in 1986 by Pr. Alain Charles Masquelet et al. IMT is a two-stage surgical operation that recently provides a more popular option for the treatment of critical size bone defect as well as fracture nonunion. Basically, first stage of IMT comprises the implantation of a polymethylmethacrylate (PMMA) cement spacer loaded with antibiotics into defect site. During 6 to 8 weeks, this spacer induces the formation and maturation of a thin layer called induced membrane surrounding it via a foreign body immune response. In stage II, the spacer is carefully removed while keeping induced membrane at the fracture site, autologous bone graft is then performed to provoke bone healing.
  Other Names: Masquelet technique
  Arms: with induced membrane
Procedure: Bone graft (Stage II of IMT) — Bone graft is only performed in this group to provoke bone healing, as same as demonstrated in the stage II of IMT.
  Arms: without induced membrane

SUMMARY:
The goal of this clinical trial is to test the role of type H vessel and investigate the mechanism of its regulation in induced membrane created by induced membrane technique in patients with open fracture, aged between 20 and 80.

The main questions to answer are:

* Whether type H vessel will be critical for induced membrane-mediated bone healing?
* Whether type H vessel will be a biomarker for diagnosing bone healing in patients with open fracture?
* To find out a circulating indicator for type H vessel in patients with open fracture undergoing induced membrane technique.

Participants will be enrolled to collect tissues of induced membrane and blood samples to detect type H vessel and measure the biomarkers of type H vessel, investigating their correlation with the capacity of bone healing. To avoid selection bias of treatment, the grouping will be achieved by a randomized protocol qualified clinical trial center of Chang Gung Memorial Hospital to divide into with induced membrane and without induced membrane. Researchers will compare these two groups to test our hypothesis that type H vessel in important in induced membrane and their corresponding biomarkers.

DETAILED DESCRIPTION:
The masquelet technique, also called an induced membrane technique (IMT), was first introduced to treat critical size bone defect up to 25 cm in 1986 by Pr. Alain Charles Masquelet et al. IMT is a two-stage surgical operation that recently provides a more popular option for the treatment of critical size bone defect as well as fracture nonunion. Basically, the first stage of IMT comprises the implantation of a polymethylmethacrylate (PMMA) cement spacer loaded with antibiotics into defect site. During 6 to 8 weeks, this spacer induces the formation and maturation of a thin layer called induced membrane surrounding it via a foreign body immune response. In stage II, the spacer is carefully removed while keeping induced membrane at the fracture site, autologous bone graft is then performed to provoke bone healing. IMT endows several beneficial effects including the relatively simple management versus vascularized fibular grafts and no significant difference in healing time among various defect sizes. Of note, multiple surgeries and long recovery time are the difficulties still needed to be conquered in patients treated with IMT. In view of the fact that induced membrane has been considered as an indispensable component for successful union, a more detailed and comprehensive analysis of it will improve the process of IMT to ameliorate those difficulties.

The clinical study design will follow the description in Chang Gung Medical Foundation Institutional Review Board, which will be begun in the first year until reaching 15 patients for each group. Briefly, patients of open fracture will be randomly divided into two groups to reduce selection bios, comprising spacer (with induced membrane) and without spacer groups (without induced membrane). In a without spacer group (No operation of stage I), soft tissues near fracture sites with a size of 1 cm2 will be collected to be used as an appropriate control of induced membrane (1 cm2) from the spacer group (Stage I + II) at the time point of stage II of IMT. Tissues will be dissected into three parts for proteomics, metabolomics, and paraffinized section, stored at minus 80 degrees prior to experiments. The section is imperative in this project to characterize type H vessel formation and the capacity of bone healing. For this purpose, immunohistochemistry (IHC) or Immunofluorescence (IF) will be performed to measure identified proteins from proteomics results in both of soft tissues and induced membrane. The characterized markers comprising cluster of differentiation 31 (CD31) and Endomucin (Emcn) will be used to detect type H vessels. Colorimetric methods including Masson's trichrome, Alcian blue, Alizarin red S, H&E and Safranin O-Fast green can also be performed to unveil histological insights of induced membrane. In the multi-omics, tissues will be used to unveil novel targets, which will then be compared to the levels of vascular endothelial growth factor (VEGF) and osteocalcin. Furthermore, western blotting and real-time reverse transcriptase-Polymerase Chain Reaction (RT-PCR) will be performed to validate downstream regulation of the identified metabolites.

The venous blood (3ml in vacutainers with heparin) will be collected from both groups at the Department of Orthopedic Surgery, Chang Gung Memorial Hospital, Taoyuan, Taiwan. The protocol was based on a report identifying VEGF as a potential biomarker of the union in IMT. After drawing, blood will be centrifuged (1000RPM, 10min at room temperature) for 30 minutes and stored at minus 80 degrees until analysis. Blood samples from the time point of collecting induced membrane are prepared for multi-omics analysis to identify systemic markers for type H vessel or induced membrane, and VEGF and osteocalcin will be used as serum indicators for bone mass. Blood samples from all time points will be used to identify a novel biomarker for type H vessels and bone healing. As for metabolite targets, targeted methods of metabolomics will be employed to verify them in blood. The time points for collecting blood samples of stage I will be the day of surgery, the next day of surgery, and 1, 2, and 4 weeks after surgery. As for stage II, the time points will be the day of surgery, the next day of surgery, and 1, 2, 12, and 14 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Accept the informed consent form
* Age: 20 years to 80 years
* Type II and III open fracture with 2-6.5 cm defect size

Exclusion Criteria:

* Not accept the informed consent form
* Age smaller than 20 years and over 80 years
* Quit during the trial
* patients with Notifiable infectious diseases such as AIDS and hepatitis as well as cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
The participants with open fracture will be assessed by the level of type H vessel | Induced membrane will be collected at 8th weeks of IMT performing procedures of stage II.
  In each group, induced membrane and soft tissue collected at 8th weeks will be used to detect CD31 and Emcn by performing immunohistochemistry (IHC) or immunofluorescence (IF), two markers for identifying type H vessel that correlated to the capacity of bone healing. The staining will be quantified as units of intensity in values defined by software or area in pixels to assess the level of type H vessel in each participant.detecting the expression level in induced membrane and soft tissue at 8 weeks, and markers of bone healing as well as metabolites in blood of each point.
The participants with open fracture will be assessed by X-ray | Bone healing tracking will be up to 24 weeks after stage II operation.
  The defect sites in these patients will be assessed the capacity of bone healing in a time-dependent manner, by quantifying the sizes of the defects from these images and representing them as the length in centimeter (cm) or area in cm2. These results will be aggregated with the level of type H vessel to report the correlation between bone healing and type H vessel.
The participants with open fracture will be assessed the metabolic alteration | Induced membrane will be collected at 8th weeks of IMT performing procedures of stage II. Blood will be a time-dependent manner through out this study up to 32 weeks.
  Finding out a potential marker to predict the correlation mentioned above, bloods collected from patients in a time-dependent manner and tissue at 8th week will be assessed the metabolic alteration by performing analysis of Liquid chromatography-mass spectrometry (LC-MS/MS). The identified metabolites will be represented as a unit of concentration in micro molar. The levels of metabolites will also be aggregated with results of type H vessel and bone healing to report whether these identified metabolites will be a type H marker defining or predicting the capacity of bone healing.

CONTACTS AND LOCATIONS:
Overall Officials: HSU YUNG-HENG, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital

REFERENCES:
- [Result] Niikura T, Oda T, Jimbo N, Komatsu M, Oe K, Fukui T, Matsumoto T, Hayashi S, Matsushita T, Itoh T, Kuroda R. Immunohistochemical analysis revealed the expression of bone morphogenetic proteins-4, 6, 7, and 9 in human induced membrane samples treated with the Masquelet technique. J Orthop Surg Res. 2022 Jan 15;17(1):29. doi: 10.1186/s13018-022-02922-y. PMID 35033126
- [Result] Tanner MC, Boxriker S, Haubruck P, Child C, Westhauser F, Fischer C, Schmidmaier G, Moghaddam A. Expression of VEGF in Peripheral Serum Is a Possible Prognostic Factor in Bone-Regeneration via Masquelet-Technique-A Pilot Study. J Clin Med. 2021 Feb 15;10(4):776. doi: 10.3390/jcm10040776. PMID 33672081